CLINICAL TRIAL: NCT05638178
Title: The Middle Norway Corona Study - Individual and Genetic Risk Factors for COVID-19 Infection.
Brief Title: The Corona Study of Middle Norway
Acronym: CUT COVID-19
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: The Research Council of Norway (Other); Alesund Hospital (Other); Namsos Hospital (Other); Molde Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: 121891
Record Dates: First submitted 2022-11-17; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease; SARS-CoV-2 Sepsis; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma (EDTA) Plasma (Citrate) Whole blood (EDTA) PBMC (CPT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult: 18+
  Interventions: Other: No intervention
- Pediatric: Under 18
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, cohort study.

SUMMARY:
CUT COVID is a cohort study establised to collect information on patients hospitalized because or with infection by SARS-CoV-2. The cohort data includes clinical data and biological samples from multiple timepoints during hospitalization, as well as data from a followup consultation 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS CoV-2 infection

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population of Middle Norway Health Region
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Predictors of COVID-19 severity | 1 year after inclusion.
  Primary aim is to assess predictors of severe COVID disease in children and adults

CONTACTS AND LOCATIONS:
Overall Officials: Kari Risnes, MD/PhD, Principal Investigator — St. Olavs Hospital
Locations (5):
- Norway (5):
  - St. Olavs Hospital, Trondheim, MN
  - Ålesund Hospital, Ålesund, MR
  - Molde Hospital, Molde, MR
  - Levanger Hospital, Levanger, NT
  - Namsos Hospital, Namsos, NT

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided on a case-by-case basis dependent on data protection impact assessment.

REFERENCES:
- [Background] Ponsford MJ, Gkatzionis A, Walker VM, Grant AJ, Wootton RE, Moore LSP, Fatumo S, Mason AM, Zuber V, Willer C, Rasheed H, Brumpton B, Hveem K, Kristian Damas J, Davies N, Asvold BO, Solligard E, Jones S, Burgess S, Rogne T, Gill D. Cardiometabolic Traits, Sepsis, and Severe COVID-19: A Mendelian Randomization Investigation. Circulation. 2020 Nov 3;142(18):1791-1793. doi: 10.1161/CIRCULATIONAHA.120.050753. Epub 2020 Sep 23. No abstract available. PMID 32966752
- [Background] COVID-19 Host Genetics Initiative. Mapping the human genetic architecture of COVID-19. Nature. 2021 Dec;600(7889):472-477. doi: 10.1038/s41586-021-03767-x. Epub 2021 Jul 8. PMID 34237774
- [Background] Degenhardt F, Ellinghaus D, Juzenas S, Lerga-Jaso J, Wendorff M, Maya-Miles D, Uellendahl-Werth F, ElAbd H, Ruhlemann MC, Arora J, Ozer O, Lenning OB, Myhre R, Vadla MS, Wacker EM, Wienbrandt L, Blandino Ortiz A, de Salazar A, Garrido Chercoles A, Palom A, Ruiz A, Garcia-Fernandez AE, Blanco-Grau A, Mantovani A, Zanella A, Holten AR, Mayer A, Bandera A, Cherubini A, Protti A, Aghemo A, Gerussi A, Ramirez A, Braun A, Nebel A, Barreira A, Lleo A, Teles A, Kildal AB, Biondi A, Caballero-Garralda A, Ganna A, Gori A, Gluck A, Lind A, Tanck A, Hinney A, Carreras Nolla A, Fracanzani AL, Peschuck A, Cavallero A, Dyrhol-Riise AM, Ruello A, Julia A, Muscatello A, Pesenti A, Voza A, Rando-Segura A, Solier A, Schmidt A, Cortes B, Mateos B, Nafria-Jimenez B, Schaefer B, Jensen B, Bellinghausen C, Maj C, Ferrando C, de la Horra C, Quereda C, Skurk C, Thibeault C, Scollo C, Herr C, Spinner CD, Gassner C, Lange C, Hu C, Paccapelo C, Lehmann C, Angelini C, Cappadona C, Azuure C; COVICAT study group, Aachen Study (COVAS); Bianco C, Cea C, Sancho C, Hoff DAL, Galimberti D, Prati D, Haschka D, Jimenez D, Pestana D, Toapanta D, Muniz-Diaz E, Azzolini E, Sandoval E, Binatti E, Scarpini E, Helbig ET, Casalone E, Urrechaga E, Paraboschi EM, Pontali E, Reverter E, Calderon EJ, Navas E, Solligard E, Contro E, Arana-Arri E, Aziz F, Garcia F, Garcia Sanchez F, Ceriotti F, Martinelli-Boneschi F, Peyvandi F, Kurth F, Blasi F, Malvestiti F, Medrano FJ, Mesonero F, Rodriguez-Frias F, Hanses F, Muller F, Hemmrich-Stanisak G, Bellani G, Grasselli G, Pezzoli G, Costantino G, Albano G, Cardamone G, Bellelli G, Citerio G, Foti G, Lamorte G, Matullo G, Baselli G, Kurihara H, Neb H, My I, Kurth I, Hernandez I, Pink I, de Rojas I, Galvan-Femenia I, Holter JC, Afset JE, Heyckendorf J, Kassens J, Damas JK, Rybniker J, Altmuller J, Ampuero J, Martin J, Erdmann J, Banales JM, Badia JR, Dopazo J, Schneider J, Bergan J, Barretina J, Walter J, Hernandez Quero J, Goikoetxea J, Delgado J, Guerrero JM, Fazaal J, Kraft J, Schroder J, Risnes K, Banasik K, Muller KE, Gaede KI, Garcia-Etxebarria K, Tonby K, Heggelund L, Izquierdo-Sanchez L, Bettini LR, Sumoy L, Sander LE, Lippert LJ, Terranova L, Nkambule L, Knopp L, Gustad LT, Garbarino L, Santoro L, Tellez L, Roade L, Ostadreza M, Intxausti M, Kogevinas M, Riveiro-Barciela M, Berger MM, Schaefer M, Niemi MEK, Gutierrez-Stampa MA, Carrabba M, Figuera Basso ME, Valsecchi MG, Hernandez-Tejero M, Vehreschild MJGT, Manunta M, Acosta-Herrera M, D'Angio M, Baldini M, Cazzaniga M, Grimsrud MM, Cornberg M, Nothen MM, Marquie M, Castoldi M, Cordioli M, Cecconi M, D'Amato M, Augustin M, Tomasi M, Boada M, Dreher M, Seilmaier MJ, Joannidis M, Wittig M, Mazzocco M, Ciccarelli M, Rodriguez-Gandia M, Bocciolone M, Miozzo M, Imaz Ayo N, Blay N, Chueca N, Montano N, Braun N, Ludwig N, Marx N, Martinez N; Norwegian SARS-CoV-2 Study group; Cornely OA, Witzke O, Palmieri O; Pa Study Group; Faverio P, Preatoni P, Bonfanti P, Omodei P, Tentorio P, Castro P, Rodrigues PM, Espana PP, Hoffmann P, Rosenstiel P, Schommers P, Suwalski P, de Pablo R, Ferrer R, Bals R, Gualtierotti R, Gallego-Duran R, Nieto R, Carpani R, Morilla R, Badalamenti S, Haider S, Ciesek S, May S, Bombace S, Marsal S, Pigazzini S, Klein S, Pelusi S, Wilfling S, Bosari S, Volland S, Brunak S, Raychaudhuri S, Schreiber S, Heilmann-Heimbach S, Aliberti S, Ripke S, Dudman S, Wesse T, Zheng T; STORM Study group, The Humanitas Task Force, The Humanitas Gavazzeni Task Force; Bahmer T, Eggermann T, Illig T, Brenner T, Pumarola T, Feldt T, Folseraas T, Gonzalez Cejudo T, Landmesser U, Protzer U, Hehr U, Rimoldi V, Monzani V, Skogen V, Keitel V, Kopfnagel V, Friaza V, Andrade V, Moreno V, Albrecht W, Peter W, Poller W, Farre X, Yi X, Wang X, Khodamoradi Y, Karadeniz Z, Latiano A, Goerg S, Bacher P, Koehler P, Tran F, Zoller H, Schulte EC, Heidecker B, Ludwig KU, Fernandez J, Romero-Gomez M, Albillos A, Invernizzi P, Buti M, Duga S, Bujanda L, Hov JR, Lenz TL, Asselta R, de Cid R, Valenti L, Karlsen TH, Caceres M, Franke A. Detailed stratified GWAS analysis for severe COVID-19 in four European populations. Hum Mol Genet. 2022 Nov 28;31(23):3945-3966. doi: 10.1093/hmg/ddac158. PMID 35848942
- See also: Official project page in the Norwegian research information system — https://app.cristin.no/projects/show.jsf?id=2497478